CLINICAL TRIAL: NCT07064317
Title: Catheter Tip Position and Contrast Distribution Following Paravertebral Catheter Insertion: a CT Study
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Chirec (Other)
Responsible Party: Principal Investigator, Imré Van Herreweghe, Anesthesiologist, Principle Investigator, Ziekenhuis Oost-Limburg
Other Study IDs: 2024/326
Record Dates: First submitted 2025-06-26; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Patients
Keywords: Thoracic paravertebral catheter; Ultrasound-guided paravertebral block; Catheter depth; Breast cancer patient; CT imaging; Catheter tip position; Mobilization; Contrast distribution; Spread

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This retrospective study aims to assess the impact of paravertebral catheter insertion depth on the final anatomical position of the catheter tip. Another objective is to characterize the contrast distribution patterns through paravertebral catheters verified to reside within the thoracic paravertebral space.

DETAILED DESCRIPTION:
The effectiveness of a continuous thoracic paravertebral block depends on optimal catheter tip placement and adequate distribution of local anesthetic. This study evaluated the relation between the catheter insertion depth and the final anatomical position of the catheter tip. Additionally, contrast distribution patterns were assessed for catheter tips residing within the thoracic paravertebral space.

Ultrasound-guided paravertebral catheters were inserted at multiple catheter insertion depths beyond the needle tip in 31 patients undergoing breast surgery. Post-mobilization computed tomography (CT) imaging was used to determine the catheter tip location. Catheter tips with a confirmed position in the paravertebral space were further analyzed for contrast distribution.

ELIGIBILITY:
Inclusion Criteria:

* Breast surgery patients who received a paravertebral catheter at Clinique Sainte-Anne Saint Rémi, Brussels, Belgium, between January 2010 and January 2012

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received a paravertebral catheter at Clinique Sainte-Anne Saint Rémi, Brussels, Belgium, between January 2010 and January 2012.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-01-27 (Actual); Primary Completion 2012-01-25 (Actual); Study Completion 2012-01-25 (Actual)

PRIMARY OUTCOMES:
Paravertebral catheter tip position | 1 Day of breast surgery
  Postoperatively, patients underwent CT scanning with 0.1 mL of contrast dye (Iomeron, iomeprol, Bracco) to precisely determine the catheter tip position and permit adjustments if needed. Two anesthesiologists independently evaluated the CT images with regards to the insertion level, depth relative to the lamina, and catheter tip location in relation to key anatomical structures. Tip locations were defined as paravertebral or non-paravertebral. Different locations were identified for both the paravertebral and the non-paravertebral spaces.
  Paravertebral space locations:
  Anterior paravertebral: Between the anterior and posterior borders of the vertebral corpus.
  Periforaminal paravertebral: Within 1 cm of the foramen. Posterior paravertebral: From the foramen to the articular process.
  Non-paravertebral locations:
  Prevertebral: Anterior to the vertebral body. Intramuscular: Posterior to the lamina within the erector spinae muscles. Epidural and Pleural: Standard anatomical definition.

SECONDARY OUTCOMES:
Paravertebral contrast distribution | 1 Day of breast surgery
  Postoperatively, patients received a CT scan with 0.1 mL of contrast dye (Iomeron, iomeprol, Bracco) to evaluate the catheter tip position. Only patients with a catheter in the paravertebral space received a second bolus of 1 mL contrast dye and 9 mL saline 0.9%. Two anesthesiologists independently evaluated the catheter tip position across the different anatomical areas close to the paravertebral space. Additionally, the contrast distribution was assessed in the anteroposterior and craniocaudal direction of catheters with a paravertebral catheter tip position.
  Paravertebral space locations:
  Anterior paravertebral: Between the anterior and posterior borders of the vertebral corpus.
  Posterior paravertebral: From the foramen to the articular process.
  Non-paravertebral locations:
  Prevertebral: Anterior to the vertebral body. Intramuscular: Posterior to the lamina within the erector spinae muscles. Epidural, Intercostal and Pleural: Standard anatomical definitions applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Sainte-Anne Saint Rémi, Brussels, Belgium